CLINICAL TRIAL: NCT05052424
Title: Cellular and Molecular Characterization of the Immune Response in Children and Adolescents With Inflammatory Syndrome in Children (MIS-C)
Brief Title: Immun Response in Children With MIS-C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, PD Dr. Katrin Mehler, Associate Professor, University of Cologne
Other Study IDs: 21-1384
Record Dates: First submitted 2021-08-31; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: MIS-C Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with MIS-C: * Children (age <18 years) hospitalized in the Children´s University Hospital of Cologne diagnosed with MIS-C (WHO criteria)
  * Assessment of clinical data
  * Blood samples are taken before therapy and on days 1,2,5,7 und 9.
  * RNA and protein expression of cytokines and immune cell-related markers will be determined via multiplex ELISA, FACS, quantitative PCR, RNAseq, and Western blot.
  Interventions: Diagnostic Test: Analysis of cytokines and immun cell related markers

INTERVENTIONS:
Diagnostic Test: Analysis of cytokines and immun cell related markers — blood samples

SUMMARY:
Multi-system inflammatory syndrome in children (MIS-C) is a post-viral inflammatory vasculopathy of children and adolescents following Covid-19 infection. It affects one of 1000-5000 children. Latency between mild or asymptomatic Covid-19 infection and MIS-C is 4-6 weeks. The immune response in MIS-C seems to be dysregulated and different from that during acute SARS-CoV-2 infection.

The investigators are planning to investigate the immune response in children with MIS-C.

RNA and protein expression of cytokines and immune cell-related markers will be determined via multiplex ELISA, FACS, quantitative PCR, RNAseq, and Western blot.

The use of highly sensitive multiplex methods will allow for the analysis of a large number of parameters in the smallest possible amount of sample. Sample preparation and analysis will be performed in close collaboration with the Centre for Molecular Medicine Cologne (CMMC) and the Institute of Virology.

With this project the investigators hope to identify risk factors for developing MIS-C and extend the knowledge on therapeutic options for the treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MIS-C (WHO criteria)
* <18 years
* Hospitalized in the Children´s University Hospital of Cologne

Exclusion Criteria:

* no informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with MIS-C
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Immune response in MIS-C | December 2022
  .The primary outcome measure is a complex pattern of numerous molecular markers of immune response determined via multiplex ELISA, FACS, quantitative PCR, RNAseq. and Western Blot. For each child, this specific molecular immune response pattern will be determined and correlated with clinical determinants allowing for the identification of predictive factors and molecular markers useful for the management of future patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Medical Faculty, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided